CLINICAL TRIAL: NCT02210091
Title: A Phase 3 Prospective, Uncontrolled, Multicenter Study Evaluating Pharmacokinetics, Efficacy, Safety, and Immunogenicity of BAX 855 (PEGylated Full-length Recombinant FVIII) in Previously Treated Pediatric Patients With Severe Hemophilia A
Brief Title: BAX 855 Pediatric Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 261202; 2014-000742-30 (EudraCT Number)
Record Dates: First submitted 2014-07-25; First posted 2014-08-06 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; BAX 855

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- <6 years old (Experimental)
  Interventions: Biological: Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method; Biological: PEGylated Recombinant Factor VIII
- ≥6 to <12 years (Experimental)
  Interventions: Biological: Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method; Biological: PEGylated Recombinant Factor VIII

INTERVENTIONS:
Biological: Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method — Pharmacokinetic (PK) analysis of ADVATE
  Other Names: ADVATE
Biological: PEGylated Recombinant Factor VIII — Pharmacokinetic (PK) analysis of BAX 855
  Other Names: BAX 855
Biological: PEGylated Recombinant Factor VIII — Prophylaxis treatment
  Other Names: BAX 855

SUMMARY:
The study purpose is:

* To assess the incidence of FVIII inhibitory antibodies during 6 months of twice weekly prophylactic treatment with BAX 855 or 50 exposure days (EDs), whichever occurs last.
* To compare pharmacokinetic (PK) parameters to ADVATE.
* To assess hemostatic efficacy in prophylaxis and the treatment of bleeding episodes.
* To evaluate safety and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A (Factor VIII (FVIII) <1%) determined by central laboratory.
* <12 years old at the time of screening.
* Participants aged ≥6 to <12 years of age have been previously treated with plasma-derived and/or recombinant Factor VIII (rFVIII) concentrate(s) for a minimum of 150 exposure days (EDs) (based on the participant's medical records).
* Participants <6 years of age have been previously treated with plasma-derived and/or rFVIII concentrate(s) for at least 50 EDs (based on the participant's medical records).
* Participant is human immunodeficiency virus (HIV) negative; or HIV positive with stable disease and CD4+ count of ≥200 cells/mm^3, as confirmed by central laboratory.
* Participant and/or legal representative accepts prophylactic treatment over a period of 6 months.
* Participant and/or the legal representative is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

* Participant has detectable FVIII inhibitory antibodies (≥0.4 Bethesda Units (BU) using the Nijmegen modification of the Bethesda assay) as confirmed by central laboratory at screening.
* Participant has a history of FVIII inhibitory antibodies (≥0.4 BU using the Nijmegen modification of the Bethesda assay or ≥0.6 BU using the Bethesda assay) at any time prior to screening.
* Participant has known hypersensitivity towards mouse or hamster proteins, polyethylene glycol (PEG), or Tween 80.
* Participant has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (eg, qualitative platelet defect or von Willebrand's disease).
* Participant's platelet count is <100,000/μL.
* Participant has severe chronic hepatic dysfunction (eg, ≥5 times upper limit of normal (ULN) alanine aminotransferase (ALT), as confirmed by central laboratory at screening, or a documented international normalized ratio (INR) >1.5).
* Participant has severe renal impairment (serum creatinine >1.5 times ULN).
* Participant is scheduled to receive during the course of the study, an immunomodulating drug (eg, corticosteroid agents at a dose equivalent to hydrocortisone >10 mg/day, or α-interferon) other than anti-retroviral chemotherapy.
* Participant has current or recent (<30 days) use of other PEGylated drugs prior to study participation or is scheduled to use such drugs during study participation.
* Participant has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
* Participant has a medical, psychiatric, or cognitive illness or recreational drug/alcohol use that, in the opinion of the Investigator, would affect participant safety or compliance.
* Participant's legal representative is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study.

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2015-10-23 (Actual); Study Completion 2015-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (39):
- United States (12):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Colorado, Denver, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Cornell University, New Hyde Park, New York
  - New York Presbyterian Hospital-Weill, New York, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
- Bulgaria (3):
  - UMHAP Sveti Georgi EAD, Plovdiv
  - Specialized Hospital for Active Treatment of Oncohematological Diseases in Children, Sofia
  - Multiprofile Hospital for Active Treatment "Sveta Marina", Varna
- The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong
- Malaysia (5):
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Hospital Sibu, Sibu, Sarawak
  - Ampang Hospital, Ampang, Selangor
  - Tengku Ampian Rahimah (TAR) Hospital, Klang, Selangor
- Academic Medical Centre, Amsterdam, Netherlands
- South Korea (3):
  - Eulji University Hosptial, Seo-gu, Daejeon
  - Ulsan University Hosptial, Dong-gu, Ulsan
  - Severance Hospital, Seoul
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Fe, Valencia
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung, Xitun District
  - China Medical University Hospital, Taichung
- Turkey (Türkiye) (4):
  - Istanbul University Faculty of Medicine, Department of Pediatric Immunology, Cerrahpaşa, Istanbul
  - Ankara University Medical Faculty, Ankara
  - Akdeniz Univesity Medical Faculty, Antalya
  - Yuzuncu Yil University Medical Faculty, Van
- Institute of Blood Pathology and Transfusion Medicine of Academy of Medical Sciences of Ukraine, Lviv, Ukraine
- United Kingdom (5):
  - Birmingham Childrens Hospital NHS Trust, Birmingham
  - St. Thomas's Hospital, London
  - Great Ormond Street Hospital For Children, London
  - Royal Manchester Children's Hospital, Manchester
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Result] Mullins ES, Stasyshyn O, Alvarez-Roman MT, Osman D, Liesner R, Engl W, Sharkhawy M, Abbuehl BE. Extended half-life pegylated, full-length recombinant factor VIII for prophylaxis in children with severe haemophilia A. Haemophilia. 2017 Mar;23(2):238-246. doi: 10.1111/hae.13119. Epub 2016 Nov 27. PMID 27891721

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 52 sites participated in this study. 39 study sites enrolled participants and 13 sites were initiated but were inactive.
Pre-assignment Details: 73 participants enrolled and were screened for study participation. There were 9 screen failures. Among these, 2 participants were screen failures at first screening but entered the study later. 66 participants were dosed in the prophylactic part of the study, of whom 31 participants were also dosed in the PK part prior to prophylaxis.
Period: Overall Study
Arm/Group | <6 Years Old | 6 to <12 Years Old
Started | 32 | 34
Completed | 32 | 32
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | <6 Years Old | 6 to <12 Years Old | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.7 (1.17) | 8.1 (1.92) | 6.0 (2.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Inhibitory Antibodies to Factor VIII (FVIII)
Description: Inhibitory antibodies to FVIII were measured using the Nijmegen modification of the Bethesda assay. Incidence of an FVIII inhibitory antibody was defined as an inhibitor level ≥0.6 Bethesda units [BU].
Time Frame: After first exposure to BAX 855 until completion of study - approx. 6 months per participant.
Population: Participants in the BAX 855 Safety Analysis Set who developed an inhibitor at any time plus participants who did not develop an inhibitor, had 50 or more exposure days (EDs) to BAX 855 and had FVIII Inhibitory test results after 50 EDs.
Measure: Number; unit: participants
Groups:
- <6 Years Old: Participants < 6 years old who received at least one dose of BAX 855.
- 6 to <12 Years Old: Participants 6 to <12 years old who received at least one dose of BAX 855.
- BAX 855 Safety Analysis Set: Participants who received at least one dose of BAX 855.
Arm/Group | <6 Years Old | 6 to <12 Years Old | BAX 855 Safety Analysis Set
Number analyzed (Participants) | 29 | 28 | 57
participants | 0 | 0 | 0

2. Secondary Outcome: Annualized Bleeding Rate (ABR)
Description: The annualized bleeding rate (ABR) during the prophylaxis period was assessed based upon each individual bleeding episode, spontaneous or traumatic, recorded in the participant´s diary and/or recorded in the physician/nurse/study site notes. The annualized bleeding rate was analyzed using a generalized linear model framework assuming a negative binomial distribution with a logarithmic link function and presence or absence of target joints and age cohort as covariates and duration of the observation period in years as offset. Point estimates for the mean and 95% confidence intervals are presented.
Time Frame: During prophylaxis period of 6 months or ≥ 50 EDs, whichever occurs last
Population: Full Analysis Set: All participants who received at least 1 dose of BAX 855 in either PK or prophylaxis part of study
Measure: Mean (95% Confidence Interval); unit: bleeding episodes per year
Groups:
- <6 Years Old: Participants <6 years old who received at least one dose of BAX 855 in either the Pharmacokinetic (PK) part of the study or the prophylaxis part of the study.
- 6 to <12 Years Old: Participants 6 to <12 years old who received at least one dose of BAX 855 in either the Pharmacokinetic (PK) part of the study or the prophylaxis part of the study.
- Full Analysis Set: Participants who received at least one dose of BAX 855 in either the Pharmacokinetic (PK) part of the study or the prophylaxis part of the study.
Arm/Group | <6 Years Old | 6 to <12 Years Old | Full Analysis Set
Number analyzed (Participants) | 32 | 34 | 66
bleeding episodes per year
  Overall annualized bleeding rate | 2.37 (3.508) [1.486 to 3.778] | 3.75 (9.046) [2.429 to 5.781] | 3.04 (6.988) [2.208 to 4.186]
  Annualized rate of joint bleeds | 0.862 (2.622) [0.381 to 1.946] | 1.355 (2.590) [0.648 to 2.833] | 1.103 (2.597) [0.637 to 1.910]
  Annualized rate of target joint bleeds | 0 (0.354) [0 to NA] — NA = infinity | 0 (1.146) [0 to NA] — NA = infinity | 0 (0.865) [0 to NA] — NA = infinity
  Annualized rate of non-target joint bleeds | 0.763 (2.618) [0.299 to 1.950] | 0.998 (2.253) [0.410 to 2.430] | 0.892 (2.420) [0.466 to 1.706]
  Annualized spontaneous bleeding rate | 1.018 (2.048) [0.523 to 1.978] | 1.316 (2.467) [0.710 to 2.438] | 1.164 (2.260) [0.740 to 1.832]
  Annualized rate of injury-related bleeds | 1.628 (2.308) [0.989 to 2.679] | 2.586 (8.678) [1.639 to 4.080] | 2.089 (6.471) [1.492 to 2.925]

3. Secondary Outcome: Consumption of BAX 855: Number of Prophylactic Infusions Per Month Per Participant
Time Frame: During prophylaxis period of 6 months or ≥ 50 EDs, whichever occurs last
Population: BAX 855 Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: infusions per month
Arm/Group | <6 Years Old | 6 to <12 Years Old | BAX 855 Safety Analysis Set
Number analyzed (Participants) | 32 | 34 | 66
infusions per month | 8.07 (0.245) | 7.72 (0.974) | 7.89 (0.736)

4. Secondary Outcome: Consumption of BAX 855: Number of Prophylactic Infusions Per Year (Annualized) Per Participant
Time Frame: During prophylaxis period of 6 months or ≥ 50 EDs, whichever occurs last
Population: BAX 855 Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: infusions per year
Arm/Group | <6 Years Old | 6 to <12 Years Old | BAX 855 Safety Analysis Set
Number analyzed (Participants) | 32 | 34 | 66
infusions per year | 96.82 (2.942) | 92.61 (11.693) | 94.65 (8.834)

5. Secondary Outcome: Consumption of BAX 855: Weight-adjusted Dose of Prophylactic Infusions Per Month Per Participant
Time Frame: During prophylaxis period of 6 months or ≥ 50 EDs, whichever occurs last
Population: BAX 855 Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | <6 Years Old | 6 to <12 Years Old | BAX 855 Safety Analysis Set
Number analyzed (Participants) | 32 | 34 | 66
IU/kg | 458.93 (46.161) | 455.86 (76.101) | 457.35 (62.919)

6. Secondary Outcome: Consumption of BAX 855: Weight-adjusted Dose of Prophylactic Infusions Per Year (Annualized) Per Participant
Time Frame: During prophylaxis period of 6 months or ≥ 50 EDs, whichever occurs last
Population: BAX 855 Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | <6 Years Old | 6 to <12 Years Old | BAX 855 Safety Analysis Set
Number analyzed (Participants) | 32 | 34 | 66
IU/kg | 5507.20 (553.931) | 5470.32 (913.210) | 5488.20 (755.033)

7. Secondary Outcome: Consumption of BAX 855: Number of Infusions Per Bleeding Episode
Time Frame: During prophylaxis period of 6 months or ≥ 50 EDs, whichever occurs last
Population: Participants in the BAX 855 Safety Analysis Set who had treated bleeding episodes.
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | <6 Years Old | 6 to <12 Years Old | BAX 855 Safety Analysis Set
Number analyzed (Participants) | 15 | 19 | 34
infusions | 1.17 (0.362) | 1.40 (0.655) | 1.30 (0.551)

8. Secondary Outcome: Consumption of BAX 855: Weight-adjusted Dose Per Bleeding Episode
Time Frame: During prophylaxis period of 6 months or ≥ 50 EDs, whichever occurs last
Population: Participants in the BAX 855 Safety Analysis Set who had treated bleeding episodes.
Measure: Mean (Standard Deviation); unit: IU/kg
Units Other Than Participants: bleeding episodes
Arm/Group | <6 Years Old | 6 to <12 Years Old | BAX 855 Safety Analysis Set
Number analyzed (Participants) | 15 | 19 | 34
Number analyzed (bleeding episodes) | 25 | 45 | 70
IU/kg
  Average dose to treat bleeding episode | 52.21 (16.681) | 62.31 (38.764) | 57.85 (31.041)
  Average dose per infusion per bleeding episode | 45.58 (10.750) | 43.76 (15.304) | 44.56 (13.327)

9. Secondary Outcome: Hemostatic Efficacy Rating for Bleeding Episodes Treated With BAX 855 at Resolution of Bleed
Description: Rating Scale for Treatment of Bleeding Episodes (BEs) (4-point ordinal scale): Excellent: Full relief of pain and cessation of objective signs of bleeding (eg, swelling, tenderness, and decreased range of motion in the case of musculoskeletal hemorrhage) after a single infusion. No additional infusion required for the control of bleeding. Administration of further infusions to maintain hemostasis did not affect this scoring. Good: Definite pain relief and/or improvement in signs of bleeding after a single infusion. Possibly requires more than 1 infusion for complete resolution. Fair: Probable and/or slight relief of pain and slight improvement in signs of bleeding after single infusion. Required more than 1 infusion for complete resolution. None: No improvement or condition worsens.
Time Frame: After first exposure to BAX 855 until completion of study - approx. 6 months per participant.
Population: Participants in the Full Analysis Set who had treated bleeding episodes.
Measure: Number; unit: bleeding episodes
Units Other Than Participants: bleeding episodes
Groups:
- <6 Years Old: Participants <6 years old who received at least one dose of BAX 855.
- Full Analysis Set: Participants who received at least one dose of BAX 855.
Arm/Group | <6 Years Old | 6 to <12 Years Old | Full Analysis Set
Number analyzed (Participants) | 15 | 19 | 34
Number analyzed (bleeding episodes) | 25 | 45 | 70
bleeding episodes
  Excellent | 15 | 19 | 34
  Good | 9 | 20 | 29
  Fair | 1 | 3 | 4
  Not reported | 0 | 3 | 3

10. Secondary Outcome: Serious Adverse Events (SAEs) Possibly or Probably Related to BAX 855
Time Frame: After first exposure to BAX 855 until completion of study - approx. 6 months per participant.
Population: BAX 855 Safety Analysis Set.
Measure: Number; unit: serious adverse events
Arm/Group | <6 Years Old | 6 to <12 Years Old | BAX 855 Safety Analysis Set
Number analyzed (Participants) | 32 | 34 | 66
serious adverse events
  Investigator Assessment | 0 | 0 | 0
  Sponsor Assessment | 0 | 0 | 0

11. Secondary Outcome: Non-serious Adverse Events Possibly or Probably Related to BAX 855
Time Frame: After first exposure to BAX 855 until completion of study - approx. 6 months per participant.
Population: BAX 855 Safety Analysis Set.
Measure: Number; unit: adverse events
Arm/Group | <6 Years Old | 6 to <12 Years Old | BAX 855 Safety Analysis Set
Number analyzed (Participants) | 32 | 34 | 66
adverse events
  Investigator Assessment | 1 | 0 | 0
  Sponsor Assessment | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs: body temperature (°C), respiratory rate (breaths/min), pulse rate (beats/min), and systolic and diastolic blood pressure (mmHg). For each vital sign value that changed from normal at baseline to abnormal at any subsequent study visit, the Investigator determined if the value was clinically significant (i.e. and adverse event), or not.
Time Frame: After first exposure to BAX 855 until completion of study - approx. 6 months per participant.
Population: BAX 855 Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | <6 Years Old | 6 to <12 Years Old | BAX 855 Safety Analysis Set
Number analyzed (Participants) | 32 | 34 | 66
participants | 1 | 0 | 0

13. Secondary Outcome: Number of Clinically Significant Changes in Clinical Laboratory Parameters (Hematology, Clinical Chemistry, Lipids)
Description: The HEMATOLOGY PANEL consisted of complete blood count: hemoglobin, hematocrit, erythrocytes (ie, red blood cell count), leukocytes (ie, white blood cell count) with differential (ie, basophils, eosinophils, lymphocytes, monocytes, and neutrophils), mean corpuscular volume, mean corpuscular hemoglobin concentration, and platelet count. The CLINICAL CHEMISTRY PANEL consisted of sodium, potassium, chloride, bicarbonate, total protein, albumin, ALT, aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase, blood urea nitrogen, creatinine, and glucose. The LIPID PANEL consisted of cholesterol, very low density lipoprotein, low density lipoprotein, high density lipoprotein, and triglycerides. For each laboratory parameter value that changed from normal at baseline to abnormal at any subsequent study visit, the Investigator determined if the value was clinically significant, or not.
Time Frame: After first exposure to BAX 855 until completion of study - approx. 6 months per participant.
Population: BAX 855 Safety Analysis Set.
Measure: Number; unit: clinically significant findings
Arm/Group | <6 Years Old | 6 to <12 Years Old | BAX 855 Safety Analysis Set
Number analyzed (Participants) | 32 | 34 | 66
clinically significant findings
  Hematology-CS Rise in Eosinophils | 1 | 0 | 1
  Clin. Chemistry-CS Rise in Alkaline Phosphatase | 1 | 0 | 1

14. Secondary Outcome: Positive Post-baseline Binding Antibodies to Factor VIII (FVIII), Polyethylene Glycol-Factor VIII (PEG-FVIII), PEG and Chinese Hamster Ovary (CHO) Proteins
Description: Binding antibodies to FVIII and PEG-FVIII, as well as to PEG, were measured using enzyme-linked immunosorbent assay (ELISA). Both immunoglobulin G (IgG) and immunoglobulin M (IgM) binding antibodies for FVIII, BAX 855, and PEG were tested at each study visit. Testing for binding antibodies to CHO was performed on citrate-anti-coagulated plasma using an ELISA employing polyclonal anti-human IgG antibodies. This outcome measure includes antibodies that were transient (antibody developed after exposure to BAX 855 but not present at study termination/completion) and pre-existent (antibody originally present before exposure to BAX 855).
Time Frame: After first exposure to BAX 855 until completion of study - approx. 6 months per participant.
Population: BAX 855 Safety Analysis Set: Data not available for 1 participant in the 6 to <12 years group as participant was prematurely withdrawn from study.
Measure: Number; unit: participants
Arm/Group | <6 Years Old | 6 to <12 Years Old | BAX 855 Safety Analysis Set
Number analyzed (Participants) | 32 | 33 | 65
participants
  Positive binding IgG antibodies to FVIII | 0 | 0 | 0
  Positive binding IgM antibodies to FVIII | 0 | 0 | 0
  Positive binding IgG antibodies to PEG-FVIII | 3 | 4 | 7
  Positive binding IgM antibodies to PEG-FVIII | 0 | 0 | 0
  Positive binding IgG antibodies to PEG | 0 | 0 | 0
  Positive binding IgM antibodies to PEG | 0 | 0 | 0
  Positive binding Ig antibodies to CHO | 0 | 0 | 0

15. Secondary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration Versus Time Curve From 0 to ∞ Hours Post-infusion (AUC0-∞)
Description: The first PK infusion was ADVATE and the second PK infusion was BAX 855. All participants undergoing PK assessment had a 72-hour washout period before administration of ADVATE and BAX 855. There were 4 blood draws for PK analysis-1 pre-infusion and 3 post infusion. The timing of the infusion (morning [am] or afternoon [pm]) and the timing of Blood Draws 3 and 4 (3 groups for each blood draw) were determined at randomization. The sequence was as follows:- Blood Draw 1. within 30 minutes pre-infusion [Day 0]; PK INFUSION - am or pm [Day 0]; Blood Draw 2. 15-30 minutes post-infusion [Day 0]; Blood Draw 3. 3 groups:- 7 hours post-infusion (if am PK infusion) or 4 hours post-infusion (if pm PK infusion) [Day 0], Day 1 am or Day 1 pm; Blood Draw 4. 3 groups:- Day 2, Day 3 or Day 4. A nonlinear mixed effects model approach (population PK) was implemented to analyze PK data. A one-stage clotting assay was used as the primary assay and a chromogenic assay was used to provide supportive data.
Time Frame: (1) within 30 min pre-infusion; (2) 15-30 min post-infusion; (3) Day 0 either 4 or 7 hours post-infusion; Day 1 am; Day 1 pm; (4) Day 2; Day 3; or Day 4
Population: Pharmacokinetic (PK) Analysis Set.
Measure: Mean (Standard Deviation); unit: IU•hr/L
Groups:
- PK Analysis Set - <6 Years Old: Participants <6 years old who had been treated with at least 1 dose of ADVATE (60 ±5 IU/kg) and 1 dose of BAX 855 (60 ±5 IU/kg) in the pharmacokinetic (PK) part of the study (prior to prophylactic treatment) and had at least 1 PK concentration available for population PK and non-compartmental analysis.
- PK Analysis Set - 6 to <12 Years Old: Participants 6 to <12 years olde who had been treated with at least 1 dose of ADVATE (60 ±5 IU/kg) and 1 dose of BAX 855 (60 ±5 IU/kg) in the pharmcokinetic (PK) part of the study (prior to prophylactic treatment) and had at least 1 PK concentration available for population PK and non-compartmental analysis.
- PK Analysis Set: Participants who had been treated with at least 1 dose of ADVATE (60 ±5 IU/kg) and 1 dose of BAX 855 (60 ±5 IU/kg) in the pharmacokinetic (PK) part of the study (prior to prophylactic treatment) and had at least 1 PK concentration available for population PK and non-compartmental analysis.
Arm/Group | PK Analysis Set - <6 Years Old | PK Analysis Set - 6 to <12 Years Old | PK Analysis Set
Number analyzed (Participants) | 14 | 17 | 31
IU•hr/L
  One stage clotting assay - ADVATE | 14000 (3070) | 14400 (1800) | 14200 (2420)
  Chromogenic assay - ADVATE | 11600 (3070) | 16600 (3290) | 14400 (4040)
  One stage clotting assay - BAX 855 | 19500 (7580) | 20100 (4930) | 19800 (6160)
  Chromogenic assay - BAX 855 | 21900 (15900) | 22600 (5140) | 22300 (11200)

16. Secondary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration Versus Time Curve From 0 to ∞ Hours Post-infusion Per Dose, (AUC0-∞/Dose)
Time Frame: as for outcome 15
Population: The PK parameters were derived using a non-compartmental estimation approach using a flexible sampling design to provide point and interval estimates for summary PK parameter using a batch method. AUC/Dose is not a standard output parameter so this calculation was not done.
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 0

17. Secondary Outcome: Pharmacokinetics (PK): Mean Residence Time (MRT)
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Pharmacokinetic (PK) Analysis Set
Measure: Mean (Standard Deviation); unit: hours (hr)
Groups:
- PK Analysis Set - 6 to <12 Years Old: Participants 6 to <12 years old who had been treated with at least 1 dose of ADVATE (60 ±5 IU/kg) and 1 dose of BAX 855 (60 ±5 IU/kg) in the pharmcokinetic (PK) part of the study (prior to prophylactic treatment) and had at least 1 PK concentration available for population PK and non-compartmental analysis.
Arm/Group | PK Analysis Set - <6 Years Old | PK Analysis Set - 6 to <12 Years Old | PK Analysis Set
Number analyzed (Participants) | 14 | 17 | 31
hours (hr)
  One stage clotting assay - ADVATE | 13.3 (3.95) | 14.2 (2.64) | 13.8 (3.27)
  Chromogenic assay - ADVATE | 12.5 (2.52) | 11.6 (1.20) | 12.0 (1.93)
  One stage clotting assay - BAX 855 | 17.0 (3.51) | 17.8 (2.40) | 17.5 (2.93)
  Chromogenic assay - BAX 855 | 18.7 (12.6) | 17.2 (3.72) | 17.9 (8.76)

18. Secondary Outcome: Pharmacokinetics (PK): Clearance (CL)
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Pharmacokinetic (PK) Analysis Set
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | PK Analysis Set - <6 Years Old | PK Analysis Set - 6 to <12 Years Old | PK Analysis Set
Number analyzed (Participants) | 14 | 17 | 31
L/hr
  One stage clotting assay - ADVATE | 0.0775 (0.0132) | 0.1250 (0.04200) | 0.1030 (0.0398)
  Chromogenic assay - ADVATE | 0.0933 (0.0106) | 0.1040 (0.00875) | 0.0994 (0.0110)
  One stage clotting assay - BAX 855 | 0.0596 (0.0190) | 0.0913 (0.0276) | 0.0770 (0.0286)
  Chromogenic assay - BAX 855 | 0.0574 (0.0174) | 0.0812 (0.0248) | 0.0704 (0.0246)

19. Secondary Outcome: Pharmacokinetics (PK): Plasma Half-life (T1/2)
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Pharmacokinetic (PK) Analysis Set
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | PK Analysis Set - <6 Years Old | PK Analysis Set - 6 to <12 Years Old | PK Analysis Set
Number analyzed (Participants) | 14 | 17 | 31
hours (hr)
  One stage clotting assay - ADVATE | 9.24 (2.74) | 9.82 (1.83) | 9.56 (2.26)
  Chromogenic assay - ADVATE | 8.68 (1.75) | 8.04 (0.83) | 8.33 (1.34)
  One stage clotting assay - BAX 855 | 11.8 (2.43) | 12.4 (1.67) | 12.1 (2.03)
  Chromogenic assay - BAX 855 | 13.0 (8.74) | 11.9 (2.58) | 12.4 (6.07)

20. Secondary Outcome: Pharmacokinetics (PK): Volume of Distribution at Steady State (Vss)
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Pharmacokinetic (PK) Analysis Set
Measure: Mean (Standard Deviation); unit: litre (L)
Groups:
- PK Analysis Set <6 Years Old: Participants <6 years old who had been treated with at least 1 dose of ADVATE (60 ±5 IU/kg) and 1 dose of BAX 855 (60 ±5 IU/kg) in the pharmacokinetic (PK) part of the study (prior to prophylactic treatment) and had at least 1 PK concentration available for population PK and non-compartmental analysis.
Arm/Group | PK Analysis Set <6 Years Old | PK Analysis Set - 6 to <12 Years Old | PK Analysis Set
Number analyzed (Participants) | 14 | 17 | 31
litre (L)
  One stage clotting assay - ADVATE | 1.02 (0.302) | 1.69 (0.350) | 1.39 (0.470)
  Chromogenic assay - ADVATE | 1.14 (0.107) | 1.20 (0.0548) | 1.18 (0.0857)
  One stage clotting assay - BAX 855 | 0.97 (0.230) | 1.59 (0.343) | 1.31 (0.427)
  Chromogenic assay - BAX 855 | 0.907 (0.124) | 1.33 (0.233) | 1.14 (0.285)

21. Secondary Outcome: Pharmacokinetics (PK): Incremental Recovery (IR)
Description: The first PK infusion was ADVATE and the second PK infusion was BAX 855. All participants undergoing PK assessment had a 72-hour washout period before administration of ADVATE and BAX 855. There were 4 blood draws for PK analysis-1 pre-infusion and 3 post infusion. The timing of the infusion (morning [am] or afternoon [pm]) and the timing of Blood Draws 3 and 4 (3 groups for each blood draw) were determined at randomization. The sequence was as follows:- Blood Draw 1. within 30 minutes pre-infusion [Day 0]; PK INFUSION - am or pm [Day 0]; Blood Draw 2. 15-30 minutes post-infusion [Day 0]; Blood Draw 3. 3 groups:- 7 hours post-infusion (if am PK infusion) or 4 hours post-infusion (if pm PK infusion) [Day 0], Day 1 am or Day 1 pm; Blood Draw 4. 3 groups:- Day 2, Day 3 or Day 4. A non-compartmental model approach was implemented to analyze IR data. A one-stage clotting assay was used as the primary assay and a chromogenic assay was used to provide supportive data.
Time Frame: as for outcome 15
Population: Pharmacokinetic (PK) Analysis Set
Measure: Mean (Standard Deviation); unit: IU/dL : IU/kg
Arm/Group | PK Analysis Set - <6 Years Old | PK Analysis Set - 6 to <12 Years Old | PK Analysis Set
Number analyzed (Participants) | 14 | 17 | 31
IU/dL : IU/kg
  One stage clotting assay - ADVATE | 1.8563 (0.76004) | 1.8696 (0.25856) | 1.8636 (0.53481)
  Chromogenic assay - ADVATE | 1.7374 (0.29110) | 2.0458 (0.31739) | 1.9065 (0.33879)
  One stage clotting assay - BAX 855 | 1.8809 (0.48894) | 1.9342 (0.47451) | 1.9101 (0.47371)
  Chromogenic assay - BAX 855 | 1.8813 (0.27069) | 2.1710 (0.38472) | 2.0402 (0.36355)

22. Secondary Outcome: Pharmacokinetics (PK): Incremental Recovery (IR) of BAX 855 Over Time - One Stage Clotting Assay
Description: Pre- and post-infusion levels of Factor VIII (FVIII) following infusion of BAX 855 were used to determine IR. For participants who underwent PK evaluation, baseline IR was determined from the IR measurement used in the PK analysis. Refer to data in Outcome measure 21- "Pharmacokinetics (PK): Incremental Recovery (IR)", for the category "One stage clotting assay - BAX 855" For participants who did not undergo a PK evaluation, baseline IR was determined at the baseline visit prior to the prophylactic treatment phase and is included in this outcome measure. Category title includes number of participants [n] < 6 yrs; ≥6 to <12 yrs and the Full Analysis Set, respectively.
Time Frame: Baseline, Week 5 (or 10-15 EDs, whichever occurs last), Week 12, and Month 6 (Completion/Termination)
Population: Participants from the Full Analysis Set who provided at least data from baseline, Week 5 (or 10-15 EDs, whichever occurred last), Week 12 or Month 6
Measure: Mean (Standard Deviation); unit: IU/dL : IU/kg
Arm/Group | <6 Years Old | 6 to <12 Years Old | Full Analysis Set
Number analyzed (Participants) | 27 | 31 | 57
IU/dL : IU/kg
  Baseline [n=15, 16, 31] | 1.6889 (0.27610) | 1.7843 (0.35942) | 1.7381 (0.32017)
  Week 5 (or after 10-15 EDs) [n= 27, 30, 57] | 1.8952 (0.55483) | 1.8661 (0.49785) | 1.8799 (0.52105)
  Week 12 [n= 26, 31, 57] | 1.6818 (0.23069) | 1.9212 (0.42496) | 1.8120 (0.36738)
  Month 6 (Termination/Completion) [n=27, 28, 55] | 1.5801 (0.31568) | 1.7120 (0.36588) | 1.6472 (0.34546)

23. Secondary Outcome: Pharmacokinetics (PK): Incremental Recovery (IR) of BAX 855 Over Time - Chromogenic Assay
Description: Pre- and post-infusion levels of Factor VIII (FVIII) following infusion of BAX 855 were used to determine IR. For participants who underwent PK evaluation, baseline IR was determined from the IR measurement used in the PK analysis. Refer to data in Outcome measure 21- "Pharmacokinetics (PK): Incremental Recovery (IR)", for the category "Chromogenic assay - BAX 855" For participants who did not undergo a PK evaluation, baseline IR was determined at the baseline visit prior to the prophylactic treatment phase and is included in this outcome measure. Category title includes number of participants [n] < 6 yrs; ≥6 to <12 yrs and the Full Analysis Set, respectively.
Time Frame: Baseline, Week 5 (or 10-15 Exposure Days [EDs], whichever occurs last), Week 12, and Month 6 (Completion/Termination)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: IU/dL : IU/kg
Arm/Group | <6 Years Old | 6 to <12 Years Old | Full Analysis Set
Number analyzed (Participants) | 27 | 31 | 57
IU/dL : IU/kg
  Baseline [n= 15; 16; 31] | 1.7675 (0.34998) | 1.9334 (0.30000) | 1.8532 (0.33055)
  Week 5 (or after 10-15 EDs) [n= 27; 30; 57] | 1.9273 (0.32400) | 1.9960 (0.39258) | 1.9635 (0.36021)
  Week 12 [n= 26; 31; 57] | 1.8794 (0.24281) | 1.9869 (0.42300) | 1.9379 (0.35368)
  Month 6 (Termination/Completion) [n= 27; 28; 55] | 1.8359 (0.29188) | 2.0659 (0.45723) | 1.9530 (0.39876)

24. Post Hoc Outcome: Pharmacokinetics (PK): Plasma Half-life Ratio of BAX 855 to ADVATE
Description: This is a descriptive summary of the ratio of plasma half-life in the same subject for BAX 855 compared to ADVATE based on the final covariate model (first observation tabulation).
Time Frame: as for outcome 15
Population: Pharmacokinetic (PK) Analysis Set
Measure: Mean (Full Range); unit: hours (hr)
Arm/Group | PK Analysis Set
Number analyzed (Participants) | 31
hours (hr)
  One stage clotting assay | 1.30 [0.944 to 2.000]
  Chromogenic assay | 1.50 [0.894 to 4.810]

ADVERSE EVENTS:
Time Frame: Throughout the study period of 1 year (8-10 months per participant)
Description: AEs were continuously monitored but specifically discussed and reviewed at these time points: pre- and post-PK infusion, at the baseline visit, during prophylactic treatment at these visits: Week 5 (or 10-15 exposure days (EDs)), Week 12, Week 20 (by phone); at the study completion visit at Month 6 or after at least 50 EDs, whichever occurred last.
Groups:
- BAX 855 Safety Analysis Set: Participants who received at least 1 dose of BAX 855.
- ADVATE Received Before BAX 855: Participants who received at least 1 dose of ADVATE prior to receiving BAX 855 in the PK part of the study.
Arm/Group | BAX 855 Safety Analysis Set | ADVATE Received Before BAX 855
Serious Adverse Events (participants affected / at risk) | 3/66 | 0/31
Other Adverse Events (participants affected / at risk) | 30/66 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAX 855 Safety Analysis Set (N=66) | ADVATE Received Before BAX 855 (N=31)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0
Gastritis (Gastrointestinal disorders) | 1 (1) | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAX 855 Safety Analysis Set (N=66) | ADVATE Received Before BAX 855 (N=31)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0
Vomiting (Gastrointestinal disorders) | 5 (6) | 0
Pyrexia (General disorders) | 13 (20) | 0
Nasopharyngitis (Infections and infestations) | 5 (5) | 0
Upper Respiratory Tract Infection (Infections and infestations) | 9 (9) | 0
Headache (Nervous system disorders) | 5 (7) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxalta's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, results may not be published without prior written approval of Sponsor.